CLINICAL TRIAL: NCT00207519
Title: The Use of Liquid Meal Replacements in Conjunction With Lifestyle Intervention in Overweight Adolescents: A 12 Week Safety and Efficacy Study
Brief Title: Liquid Meal Replacements in Conjunction With Lifestyle Intervention in Overweight Adolescents
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boston Medical Center (Other)
Responsible Party: Caroline Apovian, MD, Boston Medical Center
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: H-24640
Record Dates: First submitted 2005-09-13; First posted 2005-09-21 (Estimated); Last update posted 2009-02-11 (Estimated); Status verified 2009-02

CONDITIONS: Overweight; Obesity
Keywords: overweight; obesity; adolescent
MeSH Terms: conditions — Overweight; Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Behavioral: weekly behavioral modification group
Behavioral: liquid meal replacements

SUMMARY:
In this 3-month pilot study, we will introduce to 40 adolescents "at risk for overweight" (i.e., a BMI/age >85th percentile) a structured meal plan consisting of meal replacements, fruits, vegetables, whole grains, lean protein and dairy products. We will encourage and invite at least one parent to the scheduled visits, however, no subject will be eliminated because of lack of parental involvement. In this study, we will conduct behavior modification group sessions using lessons which are structured and patterned after the suggestions documented in the LEARNÒ Program for Weight Control. Diet instruction by a registered dietitian will include the appropriate use of meal replacements for a low-fat, low-calorie meal plan. Portion sizes of all foods recommended will be reviewed and a structured meal plan will be developed by the dietitian for subjects to follow.

Subjects will return on a weekly basis for behavioral modification groups sessions in conjunction with the liquid meal replacement diet. Blood work and physical examinations will occur pre and post intervention.

DETAILED DESCRIPTION:
In this 3-month pilot study, we will introduce to 40 adolescents "at risk for overweight" (i.e., a BMI/age >85th percentile), a structured meal plan consisting of meal replacements, fruits, vegetables, whole grains, lean protein and dairy products. We will encourage and invite at least one parent to the scheduled visits, however, no subject will be eliminated because of lack of parental involvement. Parents will be encouraged to attend group sessions designed to include behavior modification, nutrition education, physical activity recommendations, and food demonstrations as a means of family support for the subject. In this study, we will conduct behavior modification group sessions using lessons which are structured and patterned after the suggestions documented in the LEARN Program for Weight Control. Diet instruction by a registered dietitian will include the appropriate use of meal replacements for a low-fat, low-calorie meal plan. Portion sizes of all foods recommended will be reviewed and a structured meal plan will be developed by the dietitian for subjects to follow. Subjects will return for 12 weekly group sessions.

For the purposes of this pilot study, mild hypertension is defined as a systolic blood pressure of >130 but <140 mm Hg and a diastolic blood pressure of >85 but <90 mm Hg. Dyslipidemia will be defined as a total cholesterol of >200 mg/dl, LDL >130 mg/dl, HDL <40 mg/dl for male subjects and <50 mg/dl for female subjects, and triacylglycerol of >150 mg/dl. Insulin resistance/diabetes shall be defined as a fasting glucose of >110 mg/dl.

Calculating Estimated Caloric Need:

Total caloric needs for subjects with a BMI >85th% for age and sex shall be calculated using the Basal Energy Expenditure multiplied by an Activity Factor (for an estimate of total energy requirements), then subtracting 250-500 calories (to achieve a 0.5 to 1 pound weight loss per week). Basal Energy Expenditure will be calculated by using the Harris-Benedict equation as follows:

Females = 655 + 4.4(wt. in lbs) + 4.3(ht. in inches) - 4.7(age in yrs) x AF Males = 66 + 6.2(wt. in lbs) +12.7(ht. in inches) - 6.8(age in yrs) x AF

Activity Factors (AF):

1.1 Restricted Activity 1.2 Sedentary (most commonly used) 1.3 Cardiovascular Activity 3x/wk

Ideal body weight is defined as:

Females = 100 lb for the first 5 ft + 5 lb for each inch over 5 ft Males = 106 lb for the first 5 ft + 6 lb for each inch over 5 ft

Subjects will be prescribed a meal plan consisting of 3 meals and 2 snacks per day. However, 2 of the 3 meals will be replaced with a liquid meal replacement which contains 220 kcal, 10 g. protein, 40 g. carbohydrate, 2.5-3 g. fat, and 5 g. dietary fiber as well as vitamin and mineral fortification. The third meal will be high in fruits, vegetables, whole grains, lean protein (30-45 g/day) and contain 600-900 kcal. Low-calorie snacks, to include additional fruit servings, will be encouraged. The meal replacements will be taken at a time the subject will be most compliant, i.e., if subject is a chronic breakfast skipper, a meal replacement will be added for the breakfast meal. All meal replacements will be provided to the subjects at no cost; subjects will complete an order form at each visit indicating flavor choices of vanilla, chocolate or strawberry for the liquid meal replacements. They will be offered the option of a meal replacement bar versus liquid meal replacement for only one of the meal replacements per day (220 kcal, 8 g. protein, 36 g. carbohydrate, 2 g. dietary fiber). These will be a choice of chocolate peanut or granola/fruit bars.

To identify and encourage dietary compliance, subjects will be provided with a food record and will be instructed to complete 3 food records per week, two week days and one weekend day, and to indicate the time of day and which type of meal replacement was consumed. This indication will be helpful in dietary instruction regarding time of day compliance is best for consuming the meal replacement. Subjects will also be instructed to return any unused meal replacements and labels from consumed meal replacements at their regularly scheduled visits as further identification of compliance to diet. A validated Youth and Adolescent Food Frequency Questionnaire or Adolescents Food Habits Checklist will be obtained at the beginning and end of the pilot study. Blood work and a physical exam will be performed pre and post intervention.

ELIGIBILITY:
Inclusion Criteria:

* BMI >85th% for age and sex
* Weight gain over the last 6 months of >5% than expected on the growth curve
* 12-17 years of age

Exclusion Criteria:

* Subjects with intolerance to dairy products (e.g., lactose intolerance) will be excluded from entering into the study.
* Subjects must not have a history of clinically significant cardiac disease, congenital heart disease, any clinically significant abnormal cardiac condition, or be known to have a clinically significantly abnormal ECG. Specifically excluded conditions include coronary artery disease, clinically significant cardiac arrhythmias, and congestive heart failure.
* Subjects must not have a history of anorexia nervosa, untreated hypothyroidism (TSH greater than 4.0 mU/L for a second generation test), malignancy, pathophysiologic or genetic syndromes associated with obesity (i.e., Cushing's syndrome, Turner's syndrome, Prader Willi syndrome), major psychiatric illness such as bi-polar disorder, ADD, major depression, bulimia, schizophrenia, or psychosis.
* Subjects may not participate in any weight management program, except for that in this study, during this pilot. Subjects may not use prescription or over-the-counter (or herbal) weight control medication during the trial.
* Subjects must not have a history of alcohol or drug addiction or substance abuse within the previous 2 years.

Ages: 12 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 40
Dates: Start 2003-04; Primary Completion 2004-08 (Actual); Study Completion 2009-01 (Actual)

PRIMARY OUTCOMES:
Outcome measures include for efficacy of intervention, height, weight, BMI, waist circumference, percent body fat, height Z-score, weight Z-score, BMI-Z score, degree of change in weight Z-score, BMI Z-score, and percent body.

SECONDARY OUTCOMES:
Include laboratory parameters such as lipids and HbA1c.

CONTACTS AND LOCATIONS:
Overall Officials: Caroline M Apovian, MD, Principal Investigator — Boston University
Locations (1):
- Boston University Medical, Boston, Massachusetts, United States

REFERENCES:
- [Background] Ogden CL, Flegal KM, Carroll MD, Johnson CL. Prevalence and trends in overweight among US children and adolescents, 1999-2000. JAMA. 2002 Oct 9;288(14):1728-32. doi: 10.1001/jama.288.14.1728. PMID 12365956
- [Background] Troiano RP, Flegal KM. Overweight children and adolescents: description, epidemiology, and demographics. Pediatrics. 1998 Mar;101(3 Pt 2):497-504. PMID 12224656
- [Background] Strauss RS, Pollack HA. Epidemic increase in childhood overweight, 1986-1998. JAMA. 2001 Dec 12;286(22):2845-8. doi: 10.1001/jama.286.22.2845. PMID 11735760
- [Background] Barlow SE, Dietz WH. Obesity evaluation and treatment: Expert Committee recommendations. The Maternal and Child Health Bureau, Health Resources and Services Administration and the Department of Health and Human Services. Pediatrics. 1998 Sep;102(3):E29. doi: 10.1542/peds.102.3.e29. PMID 9724677
- [Background] Dietz WH. Health consequences of obesity in youth: childhood predictors of adult disease. Pediatrics. 1998 Mar;101(3 Pt 2):518-25. PMID 12224658
- [Background] Fagot-Campagna A, Pettitt DJ, Engelgau MM, Burrows NR, Geiss LS, Valdez R, Beckles GL, Saaddine J, Gregg EW, Williamson DF, Narayan KM. Type 2 diabetes among North American children and adolescents: an epidemiologic review and a public health perspective. J Pediatr. 2000 May;136(5):664-72. doi: 10.1067/mpd.2000.105141. PMID 10802501
- [Background] Ebbeling CB, Pawlak DB, Ludwig DS. Childhood obesity: public-health crisis, common sense cure. Lancet. 2002 Aug 10;360(9331):473-82. doi: 10.1016/S0140-6736(02)09678-2. PMID 12241736
- [Background] Rosenbloom AL, Joe JR, Young RS, Winter WE. Emerging epidemic of type 2 diabetes in youth. Diabetes Care. 1999 Feb;22(2):345-54. doi: 10.2337/diacare.22.2.345. PMID 10333956
- [Background] Csabi G, Torok K, Jeges S, Molnar D. Presence of metabolic cardiovascular syndrome in obese children. Eur J Pediatr. 2000 Jan-Feb;159(1-2):91-4. doi: 10.1007/pl00013812. PMID 10653338
- [Background] Whitaker RC, Wright JA, Pepe MS, Seidel KD, Dietz WH. Predicting obesity in young adulthood from childhood and parental obesity. N Engl J Med. 1997 Sep 25;337(13):869-73. doi: 10.1056/NEJM199709253371301. PMID 9302300
- [Background] Strauss RS, Knight J. Influence of the home environment on the development of obesity in children. Pediatrics. 1999 Jun;103(6):e85. doi: 10.1542/peds.103.6.e85. PMID 10353982
- [Background] McDuffie JR, Calis KA, Uwaifo GI, Sebring NG, Fallon EM, Hubbard VS, Yanovski JA. Three-month tolerability of orlistat in adolescents with obesity-related comorbid conditions. Obes Res. 2002 Jul;10(7):642-50. doi: 10.1038/oby.2002.87. PMID 12105286
- [Background] McDowell MA, Briefel RR, Alaimo K, Bischof AM, Caughman CR, Carroll MD, Loria CM, Johnson CL. Energy and macronutrient intakes of persons ages 2 months and over in the United States: Third National Health and Nutrition Examination Survey, Phase 1, 1988-91. Adv Data. 1994 Oct 24;(255):1-24. No abstract available. PMID 10141689
- [Background] Devaney BL, Gordon AR, Burghardt JA. Dietary intakes of students. Am J Clin Nutr. 1995 Jan;61(1 Suppl):205S-212S. doi: 10.1093/ajcn/61.1.205S. PMID 7832167
- [Background] Krebs-Smith SM, Cook A, Subar AF, Cleveland L, Friday J, Kahle LL. Fruit and vegetable intakes of children and adolescents in the United States. Arch Pediatr Adolesc Med. 1996 Jan;150(1):81-6. doi: 10.1001/archpedi.1996.02170260085014. PMID 8542012
- [Background] Flechtner-Mors M, Ditschuneit HH, Johnson TD, Suchard MA, Adler G. Metabolic and weight loss effects of long-term dietary intervention in obese patients: four-year results. Obes Res. 2000 Aug;8(5):399-402. doi: 10.1038/oby.2000.48. PMID 10968732
- [Background] Quinn Rothacker D. Five-year self-management of weight using meal replacements: comparison with matched controls in rural Wisconsin. Nutrition. 2000 May;16(5):344-8. doi: 10.1016/s0899-9007(99)00280-4. PMID 10793302
- [Background] Ditschuneit HH, Flechtner-Mors M, Johnson TD, Adler G. Metabolic and weight-loss effects of a long-term dietary intervention in obese patients. Am J Clin Nutr. 1999 Feb;69(2):198-204. doi: 10.1093/ajcn/69.2.198. PMID 9989680
- [Background] Heber D, Ashley JM, Wang HJ, Elashoff RM. Clinical evaluation of a minimal intervention meal replacement regimen for weight reduction. J Am Coll Nutr. 1994 Dec;13(6):608-14. doi: 10.1080/07315724.1994.10718456. PMID 7706595
- [Background] McCarron DA, Oparil S, Chait A, Haynes RB, Kris-Etherton P, Stern JS, Resnick LM, Clark S, Morris CD, Hatton DC, Metz JA, McMahon M, Holcomb S, Snyder GW, Pi-Sunyer FX. Nutritional management of cardiovascular risk factors. A randomized clinical trial. Arch Intern Med. 1997 Jan 27;157(2):169-77. PMID 9009974
- [Background] Pi-Sunyer FX, Maggio CA, McCarron DA, Reusser ME, Stern JS, Haynes RB, Oparil S, Kris-Etherton P, Resnick LM, Chait A, Morris CD, Hatton DC, Metz JA, Snyder GW, Clark S, McMahon M. Multicenter randomized trial of a comprehensive prepared meal program in type 2 diabetes. Diabetes Care. 1999 Feb;22(2):191-7. doi: 10.2337/diacare.22.2.191. PMID 10333932
- [Background] Summerbell CD, Watts C, Higgins JP, Garrow JS. Randomised controlled trial of novel, simple, and well supervised weight reducing diets in outpatients. BMJ. 1998 Nov 28;317(7171):1487-9. doi: 10.1136/bmj.317.7171.1487. PMID 9831574
- [Background] Suarez FL, Zumarraga LM, Furne JK, Levitt MD. Nutritional supplements used in weight-reduction programs increase intestinal gas in persons who malabsorb lactose. J Am Diet Assoc. 2001 Dec;101(12):1447-52. doi: 10.1016/S0002-8223(01)00349-2. PMID 11762740
- [Background] Alaimo K, McDowell MA, Briefel RR, Bischof AM, Caughman CR, Loria CM, Johnson CL. Dietary intake of vitamins, minerals, and fiber of persons ages 2 months and over in the United States: Third National Health and Nutrition Examination Survey, Phase 1, 1988-91. Adv Data. 1994 Nov 14;(258):1-28. PMID 10138938
- [Background] Leighty J, Greve L, Hembrooke T, Hood K, Hughes T, O'Brien P, Warden N, Styne D. Alterations in nutrient intake in 6-10 year old, severely obese children following a 12-week family centered integrated treatment program. Pediatric Research. 2001;49:P3-758.
- [Background] Styne D, Greve L, Hembrooke T, Hood K, Hughes T, Leighty J, O'Brien P, Warden N. Anthropomorphic and biochemical results of a family centered integrated treatment program for severely obese children. Pediatric Research. 2001;49:P3-757.
- [Background] Brownell, KD. The LEARN Program for Weight Control. Dallas, TX: American Health Publishing: 1998.